CLINICAL TRIAL: NCT04661852
Title: Phase 1 Study of Cabozantinib in Combination With Topotecan-Cyclophosphamide for Patients With Relapsed Ewing Sarcoma or Osteosarcoma
Brief Title: Cabozantinib With Topotecan-Cyclophosphamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Steven DuBois, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-535
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Relapsed Ewing Sarcoma; Refractory Ewing Sarcoma; Relapsed Osteosarcoma; Refractory Osteosarcoma
Keywords: Relapsed Ewing Sarcoma; Refractory Ewing Sarcoma; Relapsed Osteosarcoma; Refractory Osteosarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Osteosarcoma | interventions — cabozantinib; Topotecan; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CABOZANTINIB WITH TOPOTECAN-CYCLOPHOSPHAMIDE (Experimental): Participants will be accrued to dose levels in cohorts of 3 using the 3 + 3 design with a combination of cabozantinib, topotecan and cyclophosphamide.
  * Each study treatment cycle lasts 21 days.
  * Participants may receive up to 17 cycles.
  * Participants will be assigned a specific dose and schedule of the study drugs determined when enrolled in the study.
  Interventions: Drug: Cabozantinib; Drug: Topotecan; Drug: Cyclophosphamide; Drug: Myeloid growth factor

INTERVENTIONS:
Drug: Cabozantinib — PO (dose and schedule based upon dose level and nomogram)
  Other Names: COMETRIQ™
Drug: Topotecan — IV, over 30 minutes (schedule based upon dose level)
  Other Names: Hycamtin®
Drug: Cyclophosphamide — IV, over 30 minutes (schedule based upon dose level)
  Other Names: Neosar®; Cytoxan®
Drug: Myeloid growth factor — subcutaneous filgrastim (daily until ANC ≥ 1,500/mm3 after nadir) or pegfilgrastim (once) must be given, with choice of agent per institutional standard or treating physician preference, starting on day 5, 6, 7 or 8 (depending upon chemotherapy timing)
  Other Names: Filgrastim; Pegfilgrastim

SUMMARY:
This research study is a clinical trial of a new combination of drugs as a possible treatment for relapsed/refractory Ewing sarcoma and/or osteosarcoma.

* The names of the drugs are:

  * Cabozantinib
  * Topotecan
  * Cyclophosphamide
* The names of the non-investigational supportive care drugs are:

  * Filgrastim, pegfilgrastim, or a related growth factor.

DETAILED DESCRIPTION:
This is a prospective, open-label, single arm, phase 1 clinical trial. A single cohort of patients with relapsed or refractory Ewing sarcoma or osteosarcoma will be enrolled and treated in a 3+3 design with a combination of cabozantinib, topotecan and cyclophosphamide.

The research study procedures include screening for eligibility and study treatment including medical tests and follow up visits.

* The names of the drugs are:

  * Cabozantinib
  * Topotecan
  * Cyclophosphamide
* The names of the non-investigational supportive care drugs are:

  * Filgrastim, pegfilgrastim, or a related growth factor.

It is expected that up to 16 people will take part in this research study.

This research study is a Phase I clinical trial, which tests the safety of an investigational drug combination and also tries to define the appropriate doses of the drugs to use for further studies. "Investigational" means that the drug combination is being studied.

The FDA (the U.S. Food and Drug Administration) has approved all medications included in this trial as a treatment for multiple types of cancers.

The combination of topotecan and cyclophosphamide has been used for treatment of this population. Cabozantinib has been used alone for treatment of Ewing sarcoma and osteosarcoma and shown to have an effect in some patients. This is the first time that cabozantinib will be studied in combination with topotecan and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 years and ≤ 30 years at time of enrollment. Note the requirement to swallow intact pills and BSA requirement immediately following.
* BSA ≥1.25m2 and <2m2 is required.

  * Patients with BSA < 1.25m2 are not eligible for enrollment due to percent deviation of daily cabozantinib dose being too extreme as a result of limitations in the size of dose forms available.
  * Patients with BSA >2m2 are not eligible for enrollment due to inability to provide sufficient dose escalation and de-escalation for cabozantinib due to restraints imposed by dose of individual pills.
* Karnofsky performance status ≥ 50% for patients ≥16 years of age and Lansky ≥ 50% for patients <16 years of age
* Disease Requirement: Participants must have relapsed or refractory Ewing sarcoma or osteosarcoma as follows:

  * For osteosarcoma, disease must be designated as a high-grade lesion (HGOS). Diagnosis of low-grade osteosarcoma (LGOS) and parosteal osteosarcoma (POS) are excluded.
  * Histologic diagnosis consistent with Ewing sarcoma or PNET with molecular evidence of translocation involving EWSR1 or FUS (also known as TLS), such as FISH, RT-PCR, or next generation sequencing. If the translocation partner is known, it must be of the ETS family (e.g.. FLI1 or ERG). For patients referred to the study center from outside institutions, the local institutional analysis of prior tumor material may serve to fulfill this requirement.
* Patients must have fully recovered (Common Terminology Criteria for Adverse Events [CTCAE] version 5 Grade ≤1) from the acute toxic effects of all prior anti-cancer therapy except organ function. Patients must meet the following minimum washout periods prior to enrollment:
* Myelosuppressive chemotherapy

  * ≥ 14 days since the last dose of myelosuppressive chemotherapy (≥ 42 days since the last dose of nitrosourea or mitomycin C);
  * Prior use of topotecan or cyclophosphamide is permitted. Patients treated with the combination of topotecan and cyclophosphamide must meet these additional criteria:

    * No progression on the combination of topotecan/cyclophosphamide.
    * If topotecan/cyclophosphamide is the regimen immediately preceding enrollment to this trial, then no more than two prior cycles prior to transitioning to this trial.
* Radiotherapy

  * ≥ 14 days after local palliative XRT (small port);
  * ≥ 90 days after craniospinal XRT or if >50% radiation of pelvis;
  * ≥ 42 days after other substantial bone marrow radiation, including radionuclide therapy.
* Small molecule biologic therapy

  * ≥ 7 days following the last dose of a small molecule biologic agent.

    --- For agents with known adverse events occurring beyond 7 days, this duration must be extended beyond the time in which adverse events are known to occur and this should be discussed and approved by the overall PI.
  * Prior use of cabozantinib is not allowed.
  * Prior use of tyrosine kinase inhibitors (TKI), other than cabozantinib, is allowed.
* Monoclonal antibody: ≥ 21 days must have elapsed after the last dose of antibody.
* Myeloid growth factors

  * ≥ 14 days following the last dose of long-acting growth factor (e.g., pegfilgrastim);
  * ≥ 7 days following short-acting growth factor (e.g., filgrastim).
* Immunotherapy: ≥ 4 weeks since the completion of immunotherapy (e.g. tumor vaccines) aside from monoclonal antibodies with immune effects.
* Cellular therapies (e.g. CAR-T, NK or autologous stem cell boost): ≥ 42 days must have elapsed after cellular therapy.
* Wound healing & surgery

  * Patients with unhealed and/or chronic wounds are not eligible.
  * Patients with unhealed fractures are not eligible.
  * Patients must be ≥ 2 weeks from prior major surgical procedure.
  * Note: Biopsy and central line placement/removal are not considered major surgery.
* Participants must have normal organ function as defined below.

  * Hematologic requirements for subjects without known bone marrow involvement by disease:

    * Absolute neutrophil count >1000/uL
    * Platelets ≥100,000/uL and transfusion independent, defined as not receiving a platelet transfusion for at least 7 days prior to CBC documenting eligibility.
  * Hematologic requirements for subjects with bone marrow involvement by disease as demonstrated on clinically-indicated bone marrow biopsy:

    * Absolute neutrophil count >750/uL
    * Platelets ≥50,000/uL and transfusion independent, defined as not receiving a platelet transfusion for at least 7 days prior to CBC documenting eligibility.
    * Not known to be refractory to platelet or red cell transfusions.
  * Hepatic Function:

    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age (Patients with Gilbert's syndrome with a total bilirubin < 2 x ULN for age and a direct bilirubin within normal limits are permitted.
    * ALT (SGPT) ≤ 135 U/L. For the purpose of this study, the ULN for ALT is 45 U/L
    * AST ≤ 90 U/L. For the purpose of this study, the ULN for AST is 40 U/L
    * Serum albumin > 2 g/dL
  * Renal Function:

    * Serum creatinine based on age/sex as follows: Maximum Serum Creatinine (mg/dL)

      * Age 6 to < 10 years Male: 1 Female: 1
      * Age 10 to < 13 years Male: 1.2 Female1.2
      * Age 13 to < 16 years Male: 1.5 Female:1.4
      * Age ≥ 16 years Male: 1.7 Female: 1.4
      * OR Creatinine clearance ≥ 60 mL/min/1.73 m2 as obtained by nuclear medicine GFR testing for participants with creatinine levels greater than the above age/sex maximum allowed values.
    * Proteinuria: Urinalysis with urine protein < 1+ or < 1.0g/24hrs on 24-hour urine collection analysis
* Adequate Cardiac Function

  * No history of congenital prolonged QTc syndrome, NYHA Class III or IV congestive heart failure (CHF).
  * No clinically significant cardiac arrhythmias, stroke or myocardial infarction within 6 months prior to enrollment.
  * QTc ≤ 480 msec. Note: Patients with Grade 1 prolonged QTc (450-480 msec) at the time of study enrollment should have correctable causes of prolonged QTc addressed if possible (i.e., electrolytes, medications).
  * Shortening fraction of > 27% or ejection fraction of > 50% (while not receiving medications for cardiac function).
  * Adequate Blood Pressure (BP) Control, defined as:

    * For patients < 18 years old, ≤ 95th percentile for age, height and sex
    * For patients ≥ 18 years old, ≤ 140/90 mmHg
  * BP should be measured as and patients should not be receiving medication for treatment of hypertension.
* Central Nervous System Function, defined as: Patients with a known seizure disorder who are receiving non-enzyme inducing anticonvulsants and have well-controlled seizures may be enrolled.
* Adequate Coagulation, defined as: INR ≤ 1.5
* Adequate Pancreatic Function, defined as: Serum lipase ≤ 1.5 x ULN
* Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, using an institutionally approved informed consent procedure

Exclusion Criteria:

* Prior solid organ or allogeneic hematopoietic cell transplantation.
* Patients with primary or metastatic CNS Ewing sarcoma or osteosarcoma except patients with a history of CNS metastatic disease that has been resected and/or radiated without evidence of active CNS disease for 3 months preceding enrollment.
* Prohibited Concomitant Medications

  * Corticosteroids: Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, ≥ 14 days must have elapsed since last dose of corticosteroid.
  * Anti-hypertensive Medications: Patients who are currently receiving any maintenance or PRN anti-hypertensive medication are not eligible for study enrollment.
  * Investigational Drugs: Patients who are currently receiving an investigational drug are not eligible.
  * Concomitant anticoagulation with anticoagulants (e.g., warfarin, direct thrombin, Factor Xa inhibitors, heparins) or platelet inhibitors (e.g., clopidogrel, aspirin) is prohibited.
  * CYP3A4 active agents: specific CYP3A inducers and inhibitors, including enzyme-inducing anticonvulsants, are prohibited and are listed in Appendix B. They must not be taken within 7 days of starting cabozantinib.
  * QT prolonging agents: specific QT prolonging agents are prohibited. They must not be taken at the time of enrollment.
* Pregnant participants will not be entered on this study given that the effects of cabozantinib on the developing human fetus are unknown. Female participants of childbearing potential must have a documented negative pregnancy test during screening.
* Breastfeeding mothers are not eligible due to unknown risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib.
* Intercurrent illness including, but not limited to, ongoing/persistent infection (fevers >38.5 for ≥ 5 days), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a known history of HIV and/or hepatitis B (testing not required as part of screening).
* Patients with gastrointestinal disease or disorder that could interfere with absorption of cabozantinib such as bowel obstruction or inflammatory bowel disease.
* Bleeding or thrombosis:

  * Current evidence of active bleeding, intratumoral hemorrhage or bleeding diathesis.
  * Within 6 months prior to study enrollment, having history of pulmonary embolism, DVT, or other venous thromboembolic event.
  * Within 6 months prior to study enrollment, having history of significant GI bleeding, GI perforation, intra-abdominal abscess or fistula.
  * Within 6 weeks prior to study enrollment, having history of hemoptysis.
  * Within 28 days prior to study enrollment, having history of significant traumatic brain injury.
* Patients who are unable to swallow intact tablets are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerate Dose | 1 Year
  Combination of cabozantinib with cyclophosphamide and topotecan
  * If no Dose Limiting Toxicities occur during the first cycle for all three subjects, dose escalation to the next highest dose level will occur for the next three enrolling patients.
  * If one out of three patients experience a DLT during the first cycle of therapy, up to three additional subjects will then be enrolled at the same dose level for a total of six patients at this dose level. If two or more patients experience DLTs in the 1st cycle, the trial will stop enrollment and this dose level will be the MAD.
  * Up to six additional patients will be enrolled at the dose level below the MAD, with the MTD being established once ≤1 patient in a dose level experiences DLTs.
  * If two out of three patients experience DLTs during the 1st cycle, the protocol will halt enrollment at this dose level, which will be considered the MAD.

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | 1 year
  The CTCAE version 5.0 of the National Cancer Institute (NCI) for toxicity and performance reporting. Tabulations will be generated by toxicity type and grade, counting only the maximum grade per type within a given patient. Serious adverse events will be separately tabulated. This analysis will be conducted within the safety population.
Objective Response Rate | 1 year
  The objective response rate to cabozantinib, topotecan and cyclophosphamide will be calculated as follows: (# responders) / (# of patients in the response analysis population) * 100%. A 95% exact two-sided confidence interval will be placed on this proportion. In addition, the number and proportion of patients by level of response will be presented. Patients with an overall best objective response of partial response or complete response prior to local measures will be categorized as responders, and all other patients as non-responders. This analysis will be conducted within the response analysis population.
Progression Free Survival | study entry to first episode of disease progression or death, with patients without these events censored at last follow-up up to 1 year
  PFS will be estimated using Kaplan-Meier methods as time from study entry to first episode of disease progression or death, with patients without these events censored at last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C DuBois, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu